CLINICAL TRIAL: NCT05242159
Title: Prevalence and Clinical Significance of Anti-annexin A2 Antibodies in COVID-19 Infection
Acronym: IMMUNOCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0120
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19; annexin A2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In January 2020, researchers isolated and sequenced in China from patients with severe atypical pneumonia a novel coronavirus called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Coronavirus disease 2019 (COVID-19) caused by SARS-CoV-2 has rapidly spread throughout the world. SARS-CoV-2 may trigger hyperstimulation of immune system with an autoinflammatory response but also the development of an autoimmune process. These autoimmune responses may also develop through the molecular mimicry between virus and human-self components. Multiple autoantibodies have been described in COVID-19 patients.

Annexin A2 (ANXA2), an endothelial cell receptor for plasminogen and tissue plasminogen activator has been identified as a new autoantigen in antiphospholipid syndrome. ANXA2 has been identified as candidate autoantigen recognized by SARS patient sera. ANXA2 contributes also to pulmonary microvascular integrity. These data lead to identify anti-ANXA2 antibodies in COVID-19 patient sera and to know if the presence of these antibodies is associated with pulmonary injury or thrombosis in COVID-19 and represents a marker of severity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* All patients hospitalized in Amiens University Hospital with COVID-19 infection

Exclusion Criteria:

* Autoimmune diseases
* Chronic viral infection by hepatitis B virus, hepatitis C virus or human immunodeficiency virus (HIV)
* Immunosuppressive treatment
* Solid tumors
* Hematological malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in Amiens University Hospital with COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anti-ANXA2 antibodies in patients with COVID-19 infection | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France